CLINICAL TRIAL: NCT03127254
Title: Can Making Video Narratives Benefit Adolescents With Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research cancelled
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: MetroHealth Medical Center (Other); Palo Alto University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE12Z16
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Pediatric Cancer
Keywords: Video Narrative
MeSH Terms: conditions — Neoplasms | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video Narrative with surveys (Experimental): Participants will be asked to create a 10-15 minute video narrative on their experiences after being diagnosed with cancer. Participants will also be asked to complete surveys including pediatric quality of life (PedsQL), Ten Item Personality Inventory (TIPI), Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test, and The Cognitive Log (Cog-Log)
  Interventions: Behavioral: Video narrative; Behavioral: PedsQL; Behavioral: Ten Item Personality Inventory; Behavioral: Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test; Behavioral: The Cognitive Log

INTERVENTIONS:
Behavioral: Video narrative — create a 10-15 minute video intervention about teen experiences after being diagnosed with cancer
Behavioral: PedsQL — A generic 23-item Health Related Quality of Life measure initially developed using pediatric cancer patients
  Other Names: Pediatric quality of life
Behavioral: Ten Item Personality Inventory — The TIPI consists of ten items and measures personality based the subject's agreement of descriptions of themselves taken from the Big-5 model of personality
  Other Names: TIPI
Behavioral: Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test — The D-KEFS Verbal Fluency Test consists of three subtests, which take approximately 6 minutes to complete
Behavioral: The Cognitive Log — The Cog-Log is a 5-10 minute assessment designed to measure basic cognitive functioning and orientation
  Other Names: Cog-Log

SUMMARY:
The purpose of this study is to learn more about the content of and benefits of making video testimonials in adolescents with cancer.

DETAILED DESCRIPTION:
The current research aims to:

A. enlist teens with cancer to produce video narratives about their experiences with their illness B. explicitly characterize and investigate the videos' content and C. determine what aspects of the production were helpful to the teen making them and predicted to be helpful to those watching them.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer
* Patients receiving cancer treatment for the first time
* Can complete study before high school graduation
* Must be able to read and understand English

Exclusion Criteria:

* Participants cannot have been treated for other chronic illnesses prior to cancer diagnosis
* Patients with cognitive and.or verbal capacities impaired to the point where they cannot consent or assent for themselves
* Patients who cannot communicate narratives clearly due to cognitive and/or verbal impairments

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
linear regression of pediatric quality of life (PedsQL), TIPI, and coded themes from video narratives on coherence, subjectivity and redemption | at end of intervention - Approximately 60 minutes after enrolling on study
  Participants' composite scores of the 10 items that make up the emotional and social domains from the PedsQL, 15 items from the PedsQL cancer module, and the two items on the TIPI that measure Extroversion will positively covary with the resilient qualities of their narrative as measured by levels of narrative coherence, subjectivity, and redemption

SECONDARY OUTCOMES:
linear regression of coded resilient qualities of narrative with Post Video Impression Questionnaire | at end of intervention - Approximately 60 minutes after enrolling on study
  Resilient qualities of the narrative, as measured by levels of narrative coherence, subjectivity, and redemption, will predict the sum of 16 select items on the Post Video Impressions Questionnaire identifying positive impact associated with producing the narrative
linear regression of impact experienced from making the video narrative with summed scores of participants willingness to post online | at end of intervention - Approximately 60 minutes after enrolling on study
  The sum of the 16 item composite scale measuring impact experienced from making the testimonial video, on the Post Video Impressions Questionnaire, will positively predict the summed scores of two items measuring participants' willingness to post the video online
linear regression of perceived impact with summed scores of participants willingness to post the video online | at end of intervention - Approximately 60 minutes after enrolling on study
  The sum of the 7 item composite scale measuring the perceived impact on others who watch the video, on the Post Video Impressions Questionnaire, will positively predict the summed scores of two items measuring participants' willingness to post the video online

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Anderson, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center